CLINICAL TRIAL: NCT06731309
Title: ABSCESS DRAINAGE in HIDRADENITIS SUPPURATIVA: INCISION and DRAINAGE VERSUS PUNCH DEBRIDEMENT
Brief Title: HS ABSCESSES: I&D VS PUNCH DEBRIDEMENT
Acronym: HSPUNCH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Hessel H van der Zee, MD, PhD, MD, PhD, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMCD_12304
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Hidradenitis Suppurativa (Acne Inversa)
Keywords: punch biopsy tool; drainage; abscess; I&D
MeSH Terms: conditions — Hidradenitis Suppurativa; Abscess | interventions — Drainage

STUDY DESIGN:
Intervention Model Description: RCT with two intervention groups, one of which is gold standard intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Punch Debdridement (Experimental): After local anesthesia, a punch biopsy tool is positioned over the inflamed follicular unit, and a small circle of skin (4 to 8 mm in diameter) is excised. A firm twisting motion is necessary to ensure adequately deep excision. Similar to I&D, this is followed by applying digital pressure and gauze scraping to eliminate the fluid contents. The wound is then left open to allow free drainage and heal by secondary intention.
  Interventions: Procedure: Punch Debridement
- Gold standard: Incision and Drainage (Active Comparator): Incision and Drainage is a minimally invasive surgical procedure often employed for the treatment of intensely painful, tense, and fluctuant abscesses that are too deep to drain spontaneously. After administration of a broad circumferential local anesthetic, a small linear incision is made using a standard scalpel blade. Digital pressure is applied to expel the fluid collection. Saline rinses can be used to flush out the remaining contents. This method offers instant pain relief, commonly performed in acute settings by dermatologists, emergency department physicians and general practitioners.
  Interventions: Procedure: Incision and Drainage

INTERVENTIONS:
Procedure: Punch Debridement — A punch biopsy tool is positioned over the inflamed follicular unit, and a small circle of skin (4 to 8 mm in diameter) is excised. A firm twisting motion is necessary to ensure adequately deep excision.
  Arms: Punch Debdridement
Procedure: Incision and Drainage — Incision and Drainage is a minimally invasive surgical procedure often employed for the treatment of intensely painful, tense, and fluctuant abscesses that are too deep to drain spontaneously. After administration of a broad circumferential local anesthetic, a small linear incision is made using a standard scalpel blade. Digital pressure is applied to expel the fluid collection. Saline rinses can be used to flush out the remaining contents. This method offers instant pain relief, commonly performed in acute settings by dermatologists, emergency department physicians and general practitioners
  Arms: Gold standard: Incision and Drainage

SUMMARY:
This randomized-control trial is designed to determine the recurrence rate of HS abscesses following drainage via two methods: I&D with a linear incision and PD with an 8mm punch biopsy. In this context, recurrence is a newly described HS abscess adjacent to or within the previously operated area, for which a second intervention is deemed necessary. We hypothesize that PD may yield a more favorable recurrence rate. In addition to comparing recurrence rates, this randomized-control trial will also evaluate postprocedural pain, the occurrence and type of complications, and patients' quality of life associated with both procedures. These additional factors are crucial in assessing the overall effectiveness and patient satisfaction associated with each method, further informing the potential establishment of PD as the new gold standard for draining small, painful, acute HS abscesses.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with HS
* Has an abscess requiring drainage with a maximum diameter of 5 centimeters.
* Age 16 years or older
* Willing and able to provide informed consent

Exclusion Criteria:

* Has other conditions that could interfere with the study, as estimated by physician
* Unable to comply with follow-up visits
* Allergic to lidocaine and/or adrenaline.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Recurrence | 1 month
  Recurrence rate in percentage of abscesses recurring after drainage

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided